CLINICAL TRIAL: NCT04541199
Title: Randomized Crossover Trial to Compare Driving Pressures in a Closed-loop and a Conventional Mechanical Ventilation Mode in Pediatric Patients
Brief Title: Driving Pressures in a Closed-loop and a Conventional Mechanical Ventilation Mode
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Hasan ağın, Professor doctor, Head of pediatric intensive care unit (PICU), Dr. Behcet Uz Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 02018/205
Record Dates: First submitted 2020-08-24; First posted 2020-09-09 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Acute Lung Injury
Keywords: Driving pressure,; Pediatric acute respiratory distress syndrome (PARDS),; Acute lung injury (ALI),; Closed loop ventilation; Pediatric intnsive care unit (PICU)
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator)
  Interventions: Device: conventional
- Closed-loop (Experimental)
  Interventions: Device: closed loop

INTERVENTIONS:
Device: closed loop — RR and VT will be selected according to the respiratory mechanics by closed loop algorithm
  Arms: Closed-loop
Device: conventional — RR, VT, Ti will be selected by the clinician according to the respiratory mechanics
  Arms: Conventional

SUMMARY:
In mechanically ventilated patients, driving pressure (ΔP) assess the strain applied to the respiratory system and is related to ICU mortality. The aim of this randomized cross-over trial was to compare ΔP selected by a closed-loop system and by physician tailored mechanical ventilation mode. Pediatric patients admitted to PICU will be enrolled if they were invasively ventilated without any detectable respiratory effort, hemodynamic instability, or significant leakages. Two 60 minute periods of ventilation determined by randomization in APV-CMV and ASV 1.1 will be compared. Settings were adjusted to reach the same minute ventilation in both modes. ΔP will be calculated as the difference between plateau pressure and total PEEP measured using end-inspiratory and end-expiratory occlusion maneuvers, respectively.

DETAILED DESCRIPTION:
In 2015, Pediatric Acute Lung Injury Consensus Conference (PALICC) determined the pediatric acute respiratory distress syndrome (PARDS) definition. PALICC recommends using patient-specific tidal volume (VT) according to disease severity. Moreover, in the absence of transpulmonary pressure measurements (PL), an inspiratory plateau pressure limit of 28 cm H2O is recommended, allowing for slightly higher plateau pressures (29-32 cm H2O) for patients with reduced chest wall compliance. In adult ARDS, Amato et al. normalized VT to the compliance(C) by using driving pressure (ΔP) and reported that ΔP was the ventilation variable that best-stratified risk. Changes in ventilator settings resulting in a decrease in ΔP were associated with increased survival. One of the most common modes used in pediatric ventilation nowadays is synchronized controlled mandatory ventilation with adaptive pressure ventilation (APV-CMV). As compared to pressure control mode (P-CMV), APV-CMV prevents low or high VT when the compliance changes by adjusting the applied pressure. Adaptive support ventilation (ASV) is closed-loop ventilation mode, which for a given minute volume set by the clinician, adapts tidal volume (VT) and respiratory rate (RR) according to the patient's respiratory mechanics.

This prospective randomized cross over study aimed to compare ΔP between physician tailored APV-CMV mode and ASV 1.1 in pediatric mechanically ventilated patients with acute respiratory failure. After the enrollment, the patients' ventilation periods will be determined by randomization using sealed opaque envelopes. The minute ventilation, fraction of inspired O2 (FiO2) and positive end-expiratory pressure (PEEP) set by the clinician before study inclusion will be kept unchanged during all study periods. Patients will be ventilated in each mode for 60 minutes. Three consecutive -inspiratory and end-expiratory occlusion will be performed at 30 and 60 min and ΔP will be calculated for each period. Arterial blood gas will be measured at the end of each period. A wash-out period of 30 min using the ventilation mode and setting before inclusion will be performed in between the two study ventilation periods. ΔP will be calculated as the difference between plateau pressure (Pplat) and total PEEP and will be averaged for each ventilation period by using the mean of the six measurements mentioned above. VT will be calculated by integration of flow measurement. Resistance will be calculated by the least-squares fitting method. The expiratory time constant (RCexp) will be derived from the volume-flow curve at 75% of the VT and corresponding flow value. Static compliance (Cstat) will be calculated as VT divided by ΔP.

The primary outcome will be ΔP. The secondary outcome will be VT, RR, Pplat, Ti, Te, Cstat, Resistance, RCexp, pH, PaO2, PaCO2 A pilot study was performed to calculate the sample size. The mean ΔP was 12.4 (±3.31) cm H2O in ASV 1.1 and 13.5 (±4.2) cm H2O in APV-CMV. By using these pilot data, and assuming the power of 0.95 and α-error of 0.05, investigators have calculated the study size as 26 patients.

ELIGIBILITY:
Inclusion Criteria:

* All the mechanically ventilated children
* between 1-months and 18-years-old
* without any detectable respiratory effort
* whose clinical condition are not foreseen to change within the next 3 hours

Exclusion Criteria:

* septic shock
* brain death diagnose,
* with a leak equal or more than 40% of the current VT,
* receiving extracorporeal membrane oxygenation (ECMO) or targeted temperature management (TTM),

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Driving pressure | at the end of period (60th minute)
  measured with an occlusion maneuver as the difference between plateau pressure (Pplat) and total PEEP

SECONDARY OUTCOMES:
Tidal Volume (VT) | continuous measurement over 1 hour
  Integrated from flow measurement
Respiratory rate (RR) | continuous measurement over 1 hour
  Number of mechanically triggered breaths by the ventilator in 60 seconds
Expiratory time constant (RCexp) | continious measurement over 1 hour
Static compliance (Cstat) | continuous measurement over 1 hour
  will be derived from volume-flow curve at 75% of the VT and corresponding flow value
Inspiratory time (Ti) | continuous measurement over 1 hour
  Time used for inspiration during each mechanically triggered breath
Expiratory time (Te) | continuous measurement over 1 hour
  Time used for expiration during each mechanically triggered breath
pH | one measurement after 1 hour
  the measure of the hydrogen ion (H-) concentration in arterial blood
PaO2 | one measurement after 1 hour
  measurement of oxygen pressure in arterial blood
PaCO2 | one measurement after 1 hour
  measurement of CO2 pressure in arterial blood

CONTACTS AND LOCATIONS:
Locations (1):
- The Health Sciences University Izmir Behçet Uz Child Health and Diseases education and research hospital, Izmir, Turkey/izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
this will be decided depending on the approval of the patients in the written informed consent

REFERENCES:
- [Background] Santschi M, Jouvet P, Leclerc F, Gauvin F, Newth CJ, Carroll CL, Flori H, Tasker RC, Rimensberger PC, Randolph AG; PALIVE Investigators; Pediatric Acute Lung Injury and Sepsis Investigators Network (PALISI); European Society of Pediatric and Neonatal Intensive Care (ESPNIC). Acute lung injury in children: therapeutic practice and feasibility of international clinical trials. Pediatr Crit Care Med. 2010 Nov;11(6):681-9. doi: 10.1097/PCC.0b013e3181d904c0. PMID 20228688
- [Background] Pediatric Acute Lung Injury Consensus Conference Group. Pediatric acute respiratory distress syndrome: consensus recommendations from the Pediatric Acute Lung Injury Consensus Conference. Pediatr Crit Care Med. 2015 Jun;16(5):428-39. doi: 10.1097/PCC.0000000000000350. PMID 25647235
- [Background] Kneyber MCJ, de Luca D, Calderini E, Jarreau PH, Javouhey E, Lopez-Herce J, Hammer J, Macrae D, Markhorst DG, Medina A, Pons-Odena M, Racca F, Wolf G, Biban P, Brierley J, Rimensberger PC; section Respiratory Failure of the European Society for Paediatric and Neonatal Intensive Care. Recommendations for mechanical ventilation of critically ill children from the Paediatric Mechanical Ventilation Consensus Conference (PEMVECC). Intensive Care Med. 2017 Dec;43(12):1764-1780. doi: 10.1007/s00134-017-4920-z. Epub 2017 Sep 22. PMID 28936698
- [Background] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Background] Imber DA, Thomas NJ, Yehya N. Association Between Tidal Volumes Adjusted for Ideal Body Weight and Outcomes in Pediatric Acute Respiratory Distress Syndrome. Pediatr Crit Care Med. 2019 Mar;20(3):e145-e153. doi: 10.1097/PCC.0000000000001846. PMID 30640889
- [Derived] Ceylan G, Topal S, Atakul G, Colak M, Soydan E, Sandal O, Sari F, Agin H. Randomized crossover trial to compare driving pressures in a closed-loop and a conventional mechanical ventilation mode in pediatric patients. Pediatr Pulmonol. 2021 Sep;56(9):3035-3043. doi: 10.1002/ppul.25561. Epub 2021 Jul 22. PMID 34293255